CLINICAL TRIAL: NCT03438877
Title: Intensive Versus Regular Dosage For Peritoneal Dialysis In Non-Hypercatabolic Acute Kidney Injury, A Multicenter Randomized Controlled Trial
Brief Title: Intensive Versus Regular Dosage For PD In AKI.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients recruited difficult.
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong Jie, Director of PD center, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDDOSE study
Record Dates: First submitted 2018-02-08; First posted 2018-02-20 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Peritoneal Dialysis; Acute Kidney Injury
Keywords: acute kidney injury; peritoneal dialysis; dosage
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group is intensive dosage of PD.
  Interventions: Procedure: Intensive dosage of PD
- Control group (Active Comparator): Control group is regular dosage of PD.
  Interventions: Procedure: Regular dosage of PD

INTERVENTIONS:
Procedure: Intensive dosage of PD — Within the first month since PD initiates, PD prescription will be adjusted to achieve the minimum target of 3.5. It's anticipated to prescribe the dosage with automatic PD (APD) or manual PD as 24-36L/day of dialysate, 1.5-2L/exchange, and 16 cycles. Anyway, it depends on the characteristics of the patients, including residual renal function, peritoneal memberane properties. The Kt/V goal will be compromised by clinical assessment for the patient, which means PD will not induce additional treatment, such as fluid infusion.
  Other Names: intensive PD
  Arms: Intervention group
Procedure: Regular dosage of PD — Within the first month since PD initiates, PD prescription will be adjusted to achieve the minimum target of 2.1. It's anticipated to prescribe the dosage with automatic PD (APD) or manual PD as 9-12L/day of dialysate, 1.5-2L/exchange, and 6 cycles. Anyway, it depends on the characteristics of the patients, including residual renal function, peritoneal memberane properties. The Kt/V goal will be compromised by clinical assessment for the patient, which means PD will not induce additional treatment, such as fluid infusion.
  Other Names: regular PD
  Arms: Control group

SUMMARY:
This is a multicenter, pilot RCT study, aiming to compare intensive dosage and regular dosage of PD for AKI patients with indications for dialysis.

Aims of the study are to:

Examine the feasibility of the study, which aims to determine the efficacy and safety of intensive PD dose for AKI patients as compared to regular PD dose.

Establish the appropriate workflow for PD treatment for AKI patients.

DETAILED DESCRIPTION:
The incidence of acute kidney injury (AKI) is rapidly increasing worldwide, which partly due to greater recognition of AKI, more exposure to various nephrotoxins and an ageing population with increased burden of non-infectious chronic disease. Intermittent hemodialysis (IHD) or continuous renal replacement therapy (CRRT) (i.e. venous-venous HD or hemofiltration) are the most-commonly modalities applied for acute kidney injury (AKI) patients in both developed and developing countries. By contrast, the use of peritoneal dialysis (PD) has been rare. There are no consensus on the ideal dosage and target of adequacy for PD in AKI. Therefore, we are to perform a multicenter, pilot RCT study, aiming to compare intensive dosage and regular dosage of PD for AKI patients with indications for dialysis. If successful, this strategy is expected to enhance the remedy rate of AKF patients, especially in developing regions/countries.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 14 years;
* Be diagnosed as AKI according to KDIGO recommendation;
* Having indications for renal replacement therapy.

Exclusion Criteria:

* Having contraindications to peritoneal dialysis;
* Functional azotemia;
* Hypercatabolic status;
* Previous CKD history (baseline eGFR<60ml/min/1.73m2 or proteinuria);
* Psychological disorder or communication barrier;
* Pregnancy;
* Refusing to receive dialysis therapy.
* receiving mechanical ventilation.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-09-29 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
Recruitment rate of the trial | From date of randomization until the randomization of last participant.
  Recruitment rate of patients screened for the trial measured by percentage.
Retention rate of the trial | From date of randomization until 90 days after the randomization of last participant
  Retention rate of included patients in the trial measured by percentage.
Adherence rate of the trial | From date of randomization until 90 days after the randomization of last participant.
  Percentage of participants adherent to the dosing regimen of PDDOSE study.
Incidence of adverse events | From date of randomization until 90 days after the randomization of last participant.
  Incidence of adverse events measured by number of events per patient-month

SECONDARY OUTCOMES:
all cause mortality | 30-day, 60-day, 90-day after the patient enrolls in the study.
  mortality due to all causes
The rate of renal recovery | 30-day, 60-day, 90-day after the patient enrolls in the study.
  We defined renal recovery as full recovery with serum creatinine decreased to below threshold or to the baseline after dialysis withdrawal . We defined partial recovery as serum creatinine decreased by 25% or more from peak concentration but remaining higher than the threshold or baseline after dialysis withdrawal. We defined failure to recover as patient still dependent on dialysis.
length of hospital stay | 90 days of the study since the patient enrolls in the study
  total days for hospital stay
Days for dialysis treatment | From date when a patient begins peritoneal dialysis until the date of dialysis withdrawal, assessed up to 90 days.
  Days for dialysis treatment, including PD and HD
Incidence of dialysis transferring | At 90 days after patient enrolls in the study
  Incidence of dialysis transferring from PD to HD
Incidence of comorbidities | At 90 days after patient enrolls in the study
  Incidence of comorbidities, including patient's new onset comorbidities and PD-associated technique comorbidities
in-hospital cost | At 90 days after patient enrolls in the study
  in-hospital cost, including expenses of examinations, treatments and manpower cost.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Dong, PhD, Principal Investigator — Peking Universiy First Hospital
Locations (7):
- China (7):
  - Renal Division and Institute of Nephrology, Peking University First Hospital, Beijing, Beijing Municipality
  - Cangzhou central hospital, Cangzhou, Hebei
  - Nanyang City Center Hospital, Nanyang, Henan
  - Pingdingshan People's Hospital No.1, Pingdingshan, Henan
  - Minda Hospital of Hubei Minzu University, Enshi, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - The People's Hospital of Chuxiong Yi Autonomous Prefecture, Chuxiong, Yunnan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cullis B, Abdelraheem M, Abrahams G, Balbi A, Cruz DN, Frishberg Y, Koch V, McCulloch M, Numanoglu A, Nourse P, Pecoits-Filho R, Ponce D, Warady B, Yeates K, Finkelstein FO. Peritoneal dialysis for acute kidney injury. Perit Dial Int. 2014 Jul-Aug;34(5):494-517. doi: 10.3747/pdi.2013.00222. No abstract available. PMID 25074995